CLINICAL TRIAL: NCT03547869
Title: Investigating Pain in Gulf War Illness With Transcranial Direct Current Stimulation.
Brief Title: Transcranial Direct Current Stimulation for Pain Treatment in Gulf War Illness.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding finished
Sponsor: The University of Texas at Dallas (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Sven Vanneste, Associate professor, The University of Texas at Dallas
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 17-88
Record Dates: First submitted 2018-03-16; First posted 2018-06-06 (Actual); Results first posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Gulf War Syndrome
Keywords: Transcranial Direct Current Stimulation; Gulf War Illness; Pain modulation
MeSH Terms: conditions — Persian Gulf Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active tDCS (Experimental): Active tDCS
  Interventions: Device: Active tDCS
- Sham tDCS (Sham Comparator): Sham tDCS
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Active tDCS — Active tDCS will be adminestered
  Arms: Active tDCS
Device: Sham tDCS — Sham tDCS will be administered
  Arms: Sham tDCS

SUMMARY:
The goal of this study is to investigate long-term modulation of pain pathways leading to a suppression of pain symptoms in Gulf War Illness patients by applying transcranial direct current stimulation.

DETAILED DESCRIPTION:
Gulf War Illness is a chronic and multisymptomatic disorder affecting returning military veterans of the 1990-1991 Gulf war. Pain is a major complaint of Gulf War Illness patients and is a leading cause of disability in veterans diagnosed with musculoskeletal ailments including joint and muscle pain, muscle fatigue, difficulty with lifting objects, and extremity paresthesia's. As a result, the target of the present study is the treatment of the pain symptoms, as this is detectable across all Gulf War Illness case classification systems.

Transcranial Direct current stimulation (tDCS) is a non-invasive and painless electrical stimulation technique that has already demonstrated to improve pain symptoms in other patient populations, e.g. fibromyalgia patients. To investigate whether we can improve pain symptoms in GWI patients with pain complaints, we will compare behavioral (questionnaires) and electrophysiological (Electroencephalography) measures before and immediately after 10 sessions of tDCS and on several follow up sessions after the last tDCS from 2 groups.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female US military veterans serving during the 1990-1991 Gulf War.
2. Men and women between the ages of 18 and 50 years old during service in the Gulf War (born between 1940 and 1973).
3. English speakers.

Exclusion Criteria:

1. Non-English speakers.
2. History of a neurological disorder, including dementia of any type, moderate to severe traumatic brain injury (TBI), brain tumors, present or past drug abuse, stroke, blood vessel abnormalities in the brain, Parkinson's disease, Huntington's disease, or multiple sclerosis. Traumatic brain injury will be screened by history.
3. No subjects will be enrolled who are cognitively or clinically incompetent to give informed consent.
4. Subjects cannot be taking medications that include: amphetamines, L-dopa, carbamazepine, sulpiride, pergolide, lorazepam, rivastigmine, dextromethorphan, D-cycloserine, flunarizine, ropinirole,or citalopram.
5. Subjects with cardiac pacemakers, implanted medication pumps of any sort, or a history of bad heart disease, a history of seizures and/or family members with a history of seizures, and/or the presence of any metal objects in or near the head which cannot be safely removed for the duration of this study.

Ages: 45 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2023-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sven Vanneste, PhD, Principal Investigator — The University of Texas at Dallas
Locations (2):
- United States (2):
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Texas at Dallas, Richardson, Texas

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active tDCS | Sham tDCS
Started | 6 | 3
Completed | 2 | 1
Not Completed | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active tDCS | Sham tDCS | Total
Number analyzed (Participants) | 6 | 3 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 3 | 9
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 3 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Pain Symptom Changes Will be Measured by a Visual Analogue Scale for Pain .
Description: Pain symptoms changes will be assessed by a Visual Analogue Scale for pain and the results will be compared between the two groups (active tDCS and sham tDCS) to study any possible differences occurring throughout the sessions.
  0 no pain - 100 cm maximum pain you can imagine.
Time Frame: Before tDCS stimulation (baseline), immediately after (immediate-post) tDCS intervention measurements and 1 week, 4 weeks, 12 weeks and 24 weeks after the last tDCS session.
Population: We had to stop collection of our data-collection due to COVID, as the IRB did not allow us to continue to collect human data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 6 | 3
score on a scale
  Baseline | 67.1 (5.35) | 68.2 (6.98)
  immediate after | 53.21 (9.10) | 63.21 (7.90)
  week 1: number analyzed (Participants) | 3 | 2
  week 1 | 54.23 (12.91) | 64.20 (13.45)
  week 4: number analyzed (Participants) | 0 | 0
  week 12: number analyzed (Participants) | 0 | 0
  week 24: number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: adverse event and/or serious adverse event, used to collect adverse event information, do not differ from the clinicaltrials.gov Definitions
Arm/Group | Active tDCS | Sham tDCS
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/3
Other Adverse Events (participants affected / at risk) | 0/6 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-06-20): https://cdn.clinicaltrials.gov/large-docs/69/NCT03547869/Prot_006.pdf
  • Statistical Analysis Plan (2017-06-20): https://cdn.clinicaltrials.gov/large-docs/69/NCT03547869/SAP_009.pdf